CLINICAL TRIAL: NCT04951466
Title: Mindfulness Based Therapy for Insomnia in Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000030653
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Insomnia
Keywords: Mindfulness-based therapy for insomnia (MBTI)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based therapy for insomnia (MBTI) (Experimental): Participants randomly assigned to the MBTI will receive 2 hours weekly session of mindfulness meditation and behavioral sleep strategies for 8 weeks.
  Interventions: Behavioral: Mindfulness-based therapy for insomnia (MBTI)
- Healthy Lifestyle Education (Active Comparator): Participants in the control group will receive sessions on the following topics: Introduction to health promotion, disease prevention and screening, healthy eating, physical activity, communication, and endings.
  Interventions: Behavioral: Healthy lifestyle intervention

INTERVENTIONS:
Behavioral: Mindfulness-based therapy for insomnia (MBTI) — Participants randomly assigned to either the MBTI or healthy lifestyle intervention will receive 2 hours weekly session of mindfulness meditation and behavioral sleep strategies for 8 weeks.
  Arms: Mindfulness-based therapy for insomnia (MBTI)
Behavioral: Healthy lifestyle intervention — Participants randomly assigned to either the MBTI or healthy lifestyle intervention will receive 2 hours weekly session of mindfulness meditation and behavioral sleep strategies for 8 weeks.
  Arms: Healthy Lifestyle Education

SUMMARY:
The purpose of the study is to conduct an 8-week RCT to improve insomnia among black women with insomnia and evaluate its feasibility, acceptability, and efficacy of Mindfulness Based Therapy for Insomnia (MBTI)

DETAILED DESCRIPTION:
Study design is a randomized clinical trial (RCT) with attention control. Participants will be randomly assigned to participate in either Mindfulness Based Therapy for Insomnia (MBTI) or time and attention control. Participants in the experimental group will receive the MBTI that includes mindfulness meditation and behavioral strategies for sleep. Participants in the control group will receive healthy lifestyle education that includes healthy eating, physical activity and sleep hygiene practice to mitigate insomnia.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Black women
* 25-45 years old
* English speaking
* meeting DSM-5/ICSD3 diagnostic criteria for insomnia disorders defined as difficulty initiating or maintaining sleep with at least one associated daytime impairment symptom (Insomnia severity index > 7)

Exclusion Criteria:

* Psychosis or unstable/ significant depression, anxiety, or substance abuse under active care (more than 1 monthly mental healthcare visit or requiring more than 1 psychotropic medicine daily)
* significant current practice of any form of meditation (>15min per day)
* obstructive sleep apnea (OSA), restless legs syndrome (RLS), or circadian rhythm related condition (shift worker, pregnancy, use of medication that influence circadian rhythm, e.g., Parkinson's disease)
* other medical conditions that confound salivary biomarkers outcomes (e.g., radiation of salivary glands, Cushing or Addison's disease)
* active or terminal cancer

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified Black women
Enrollment: 30 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Retention | 10 weeks
  Retention will be measured in the study. The following information will be collected: percentage of participants completing baseline and follow-up assessments, reasons for dropouts
Enrollment | 10 weeks
  The refusal rate of enrollment will be used to measure enrollment to determine feasibility
Change in Fidelity | Baseline and week 10
  Fidelity: Self-report checklist by interventionists and observers. We will use the Treatment Fidelity Tool for Mindfulness Interventions.
Change in Insomnia severity score | Baseline and week 10
  The reliable and valid Insomnia severity Index (ISI) for clinical diagnosis for insomnia (ICSD) will be used to determine insomnia severity score. Clinical cut points for ISI are as follows: no insomnia (0-7), sub-threshold insomnia (8-14), moderate insomnia (15-21), and severe insomnia (22-28). Response to the intervention on the ISI will be defined as a meaningful change of 7 or more points from baseline, or remission as reduction to a score less than 8.
Change in sleep onset latency | Baseline and week 10
  Sleep onset latency is the amount of time, in minutes, it takes a person to fall asleep. It begins at "light out' when the lights are turned off and the person attempts to fall asleep, and ends at sleep onset. A sleep latency of 10-20 minutes is considered normal.
Change in sleep efficiency and quality | Baseline and week 10
  Will be measured by a wrist sleep actigraphy and sleep diary. Sleep efficiency is defined by the ratio of total sleep time to time in bed. Normal sleep efficiency for a healthy adult is 90% or higher. Sleep quality will be collected by participant's self-report using a 0-10 numerical scale (higher score means better sleep quality)
Change in wake after sleep onset | Baseline and week 10
  Wake after sleep onset (WASO) is the amount of wake time in minutes during the attempted sleeping period after sleep onset has been achieved.
Change in total sleep time | Baseline and week 10
  Total sleep time or duration is computed by asking participants what time they wake-up and what time they go to bed (range from 0 min-1440 min).
Change in perceived stress score (PSS) | Baseline and week 10
  The PSS has 10 items. It measures feelings and stressful thoughts for the past month. PSS ranges from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.

SECONDARY OUTCOMES:
Change in Cortisol | Baseline and week 10
  Cortisol measures levels of salivary stress. Within-group changes, compared with control, of cortisol biomarkers outcomes will be measured. Test volume, lower limit of sensitivity, range of calibrators are as follows: 25 ul, .007 ug/dl, .012 - 3.0 ug/dl for cortisol
Change in C-reactive protein [CRP] | Baseline and week 10
  Within-group changes, compared with control, of C-reactive protein [CRP] biomarkers outcomes will be measured. Test volume, lower limit of sensitivity, range of calibrators are as follows: 100 ul, 9.72 pg/ml, 25-1600 pg/ml for CRP.
Change in cytokines [IL-1β, IL-6, TNF- α]) | Baseline and week 10
  Within-group changes, compared with control, of cytokines [IL-1β, IL-6, TNF- α]) biomarkers outcomes will be measured. Test volume, lower limit of sensitivity, range of calibrators are as follows: 60 ul, .07 pg/ml, 0-100 pg/ml for IL-6.
Change in Patient Health Questionnaire (PHQ-9) | Baseline and week 10
  PHQ-9 assesses depression symptoms. Each item asks about the frequency of specific depressive symptoms experienced over the past two weeks. The response options are scored from 0 to 3, indicating "not at all" to "nearly every day." The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms. The scoring can also be divided into categories, with scores of 0-4 indicating minimal or no depression, 5-9 indicating mild depression, 10-14 indicating moderate depression, 15-19 indicating moderately severe depression, and 20 or above indicating severe depression.
Change in The Epworth Sleepiness Scale | Baseline and week 10
  The Epworth Sleepiness Scale: measures general level of daytime sleepiness. Each question is rated on a scale of 0 to 3, with 0 indicating no chance of dozing and 3 indicating a high chance of dozing. The total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.
Change in The Dysfunctional Beliefs and Attitudes about Sleep (DBAS) | Baseline and week 10
  DBAS is a 16 item-scale evaluates the following sleep-related cognitions: consequences of insomnia, worry about sleep, sleep expectations, and medication. Each item is rated on a 10-point scale ranging from 1 (strongly disagree) to 10 (strongly agree). For each statement, participants rated their level of agreement/disagreement by choosing "strongly disagree" (0) to "strongly agree" (10). The subscale score is calculated with the average score of items. A higher score indicates more dysfunctional beliefs and attitudes about sleep.
Change in The Sleep Hygiene Practice Scale (SHPS) | Baseline and week 10
  The Sleep Hygiene Practice Scale (SHPS): assesses sleep hygiene awareness and practices. The SHPS has 19 items which include sleep-related behaviors (napping, caffeine/alcohol intake), night time activities (exercise, phone conversation), and bedroom environment (noise, light, temperature and bed partner). Respondents report on the average number of days per week in which they engaged in these activities during the previous month. Frequency scores (number of days per week) were calculated for each item, and higher frequency scores indicated worse sleep hygiene practices. The total hygiene practice scores ranged from 0 to 133.
Change in The Trait Anxiety Scale | Baseline and week 10
  The Trait Anxiety Scale consists of 20 self-report items that assess how individuals generally feel and respond to various situations in their lives. Participants are asked to rate the frequency or intensity of their anxiety-related feelings, thoughts, and behaviors on a Likert scale. The scale typically ranges from 1 to 4 or 1 to 5, with higher scores indicating higher levels of trait anxiety.
Change in Five Facet Mindfulness Questionnaire (FFMQ) | Baseline and week 10
  The Five Facet Mindfulness Questionnaire (FFMQ) will be used to measure adherence to the study protocol. The FFMQ Short Form has 24 items. Responses in the scale are made on a 5-point Likert Scale. Total FFMQ can be divided by 24 to get an average item score. The five facets, or five key aspects of mindfulness that the test measures acts as the mediator of therapeutic change and mindful interventions. Higher score means higher level in mindfulness practice.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline and week 10
  PSQI measures seven components: sleep quality, sleep latency, sleep duration, habitual sleep efficiency (percentage of total time in bed spent in sleep), sleep disturbances, use of sleep medications, and daytime dysfunction. Each component has a range from 0 (no difficulty) to 3 (severe difficulty). The global score of PSQI ranges from 0 to 21, with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University - West Campus, Orange, Connecticut, United States